CLINICAL TRIAL: NCT02742311
Title: EuroPainClinics® Study V (Prospective Observational Study)
Acronym: EPCSV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Europainclinics z.ú. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EK: 9N-2015
Record Dates: First submitted 2016-04-10; First posted 2016-04-19 (Estimated); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Back Pain; Intervertebral Disc Herniation
MeSH Terms: conditions — Back Pain; Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transforaminal endoscopic discectomy (Active Comparator)
  Interventions: Procedure: Endoscopic disectomy
- interlaminar endoscopic discectomy (Active Comparator)
  Interventions: Procedure: Endoscopic disectomy

INTERVENTIONS:
Procedure: Endoscopic disectomy — Endoscopic discectomy is an established method for treatment of lumbar disc herniation. Edoscopic discectomy provides a safe and minimal access corridor for lumbar discectomy. The technique also allows early postoperative mobilization and faster return to work.

SUMMARY:
In this prospective observational trial the effect of the Endoscopic discectomy microinvasive therapy should be examined in (approximately 500) adult patients with low back pain.

ELIGIBILITY:
Inclusion Criteria:

* lumbar disc prolapse with unilateral radiculopathy, on clinical evaluation, positive straight leg raise or femoral stretch test, and identification of a single nerve root lesion on MRI

Exclusion Criteria:

* The exlusion criteria: bilateral root symptoms, double root involvement, cauda equina syndrome and negative MRI Picture for disc herniation, unsigned infomed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2021-12-31 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
1.Pain as assessed by the Visual analogue scale All acquired information will be noted in to the special anonymous protocol | 3 years
  All acquired information will be noted in to the special anonymous protocol

SECONDARY OUTCOMES:
2.Pain localization as assessed by note of radiating dermatome as neurologic examination | 3 years
  All acquired information will be noted in to the special anonymous protocol
3.Pain progress as assessed by global pain scale | 3 years
  All acquired information will be noted in to the special anonymous protocol
4. Changes in analgesics drugs consumption as assessed by equianalgesic dose ratios for opioids | 3 years
  All acquired information will be noted in to the special anonymous protoco

CONTACTS AND LOCATIONS:
Overall Officials: Miroslav Burianek, MD MPH, Study Chair — Director
Locations (1):
- Europainclinics algesiology ambulance, Bardejov, Slovakia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rapcan R, Kocan L, Witkovsky V, Rapcanova S, Mlaka J, Tirpak R, Burianek M, Kocanova H, Vaskova J, Gajdos M. Endoscopic discectomy of the herniated intervertebral disc and changes in quality-of-life EQ-5D-5L analysis. Medicine (Baltimore). 2023 Jun 30;102(26):e34188. doi: 10.1097/MD.0000000000034188. PMID 37390280